CLINICAL TRIAL: NCT04302181
Title: Augmenting Massed Prolonged Exposure With a Stellate Ganglion Block to Treat Posttraumatic Stress Disorder (PTSD) in Active Duty or Retired Service Members: A Pilot Study
Brief Title: Augmenting Massed Prolonged Exposure With a Stellate Ganglion Block to Treat PTSD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20190878H
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: A small open-label treatment study
Masking Description: Masked clinical diagnostic assessor for the CAPS-5
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stellate Ganglion Block (Experimental): One time administration of a stellate ganglion block
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — 6.5cc of Ropivacaine HCl 0.5%, one time into the stellate ganglion
  Other Names: Naropin

SUMMARY:
This is a small, open-label treatment study that tests the potential safety and treatment effectiveness of a stellate ganglion block combined with Massed Prolonged Exposure (PE). Each of the 12 participants will receive ten 90-minute sessions of Massed Prolonged Exposure and an injection of a stellate ganglion block between the first and second PE sessions.

DETAILED DESCRIPTION:
Massed PE will be conducted by doctoral-level therapists. Participants will meet with their providers for individual, 90-minute sessions. They will then be asked to complete out-of-session treatment assignments throughout the rest of the day. Between the individual therapy session and out-of-session treatment assignments, participants will engage in approximately four to six hours of treatment per day, Monday through Friday, for two weeks. The stellate ganglion block injection will be administered between the first and second massed PE session by qualified medical personnel as per standard operating procedure for the placement of a stellate ganglion block. A research nurse will be in attendance during the procedure and for an hour recovery period following the block administration.

During PE treatment, participants will complete interim assessments of their PTSD symptoms, mood symptoms, trauma-related cognitions, and suicidal ideation proceeding sessions 6 and 10.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty or retired military service member (age 18- 65 years)
2. PTSD diagnosis as assessed by Clinician-Administered Posttraumatic Stress Scale (CAPS-5)
3. Able to speak and read English (due to standardization of outcome measures)
4. Defense Enrollment Eligibility Reporting System (DEERS)-eligible to receive care at Brooke Army Medical Center for the stellate ganglion block.

Exclusion Criteria:

1. Classification as high risk for suicide
2. Current serious mental health diagnosis (e.g., bipolar or psychosis)
3. Symptoms of moderate to severe substance (to include alcohol) use within the last 30 days
4. Pregnancy (i.e. positive pregnancy test at screening) or breastfeeding
5. Current anticoagulant use
6. History of bleeding disorder
7. Infection or mass at injection site
8. Myocardial infarction within 6 months of procedure
9. Pathologic bradycardia or irregularities of heart rate or rhythm;
10. Symptomatic hypotension
11. Phrenic or laryngeal nerve palsy
12. History of glaucoma
13. Uncontrolled seizure disorder
14. History of allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Change in CAPS-5 (Clinician-Administered PTSD Scale) | Baseline, 1 month and 3 months
  A 30-item structured interview used to assess symptoms of PTSD. Questions target the onset and duration of symptoms, subjective distress, impact on social and occupational functioning.
Change in PCL-5 (Posttraumatic Stress Disorder Checklist) | Baseline, 1 month and 3 months
  A 20-item self-report measure that assesses the presence and severity of PTSD symptoms using the Diagnostic and Statistical Manual of mental disorders (DSM-5).

SECONDARY OUTCOMES:
Change in PHQ-9 (Patient Health Questionnaire-9) | Baseline, 1 month and 3 months
  A 9-item self-report measure that assesses the presence and severity of depressive symptoms.
Change in Brief Inventory of Psychosocial Functioning | Baseline, 1 month and 3 months
  A 7-item self-report measure assessing respondents' level of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living.
Change in GAD-7 (General Anxiety Disorder Screener) | Baseline, 1 month and 3 months
  A 9-item self-report measure that assesses the presence and severity of general anxiety symptoms.
Change in PTCI (Posttraumatic Cognitions Inventory) | Baseline, 1 month and 3 months
  A 36-item self-report measure that assesses self-blame, negative cognitions about self, and negative cognitions about the world following trauma exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Peterson, PhD, ABPP, Principal Investigator — University of Texas Health San Antonio Texas at San Antonio
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foa EB, McLean CP, Zang Y, Rosenfield D, Yadin E, Yarvis JS, Mintz J, Young-McCaughan S, Borah EV, Dondanville KA, Fina BA, Hall-Clark BN, Lichner T, Litz BT, Roache J, Wright EC, Peterson AL; STRONG STAR Consortium. Effect of Prolonged Exposure Therapy Delivered Over 2 Weeks vs 8 Weeks vs Present-Centered Therapy on PTSD Symptom Severity in Military Personnel: A Randomized Clinical Trial. JAMA. 2018 Jan 23;319(4):354-364. doi: 10.1001/jama.2017.21242. PMID 29362795
- [Background] Hanling SR, Hickey A, Lesnik I, Hackworth RJ, Stedje-Larsen E, Drastal CA, McLay RN. Stellate Ganglion Block for the Treatment of Posttraumatic Stress Disorder: A Randomized, Double-Blind, Controlled Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):494-500. doi: 10.1097/AAP.0000000000000402. PMID 27187898
- [Background] Gunduz OH, Kenis-Coskun O. Ganglion blocks as a treatment of pain: current perspectives. J Pain Res. 2017 Dec 14;10:2815-2826. doi: 10.2147/JPR.S134775. eCollection 2017. PMID 29276402
- [Background] Lipov EG, Joshi JR, Lipov S, Sanders SE, Siroko MK. Cervical sympathetic blockade in a patient with post-traumatic stress disorder: a case report. Ann Clin Psychiatry. 2008 Oct-Dec;20(4):227-8. doi: 10.1080/10401230802435518. No abstract available. PMID 19034755
- [Background] Lynch JH, Mulvaney SW, Kim EH, de Leeuw JB, Schroeder MJ, Kane SF. Effect of Stellate Ganglion Block on Specific Symptom Clusters for Treatment of Post-Traumatic Stress Disorder. Mil Med. 2016 Sep;181(9):1135-41. doi: 10.7205/MILMED-D-15-00518. PMID 27612365
- [Background] Mulvaney SW, Lynch JH, Hickey MJ, Rahman-Rawlins T, Schroeder M, Kane S, Lipov E. Stellate ganglion block used to treat symptoms associated with combat-related post-traumatic stress disorder: a case series of 166 patients. Mil Med. 2014 Oct;179(10):1133-40. doi: 10.7205/MILMED-D-14-00151. PMID 25269132
- [Derived] Peterson AL, Straud CL, Young-McCaughan S, McCallin JP, Hoch M, Roux NP 3rd, Koch L, Lara-Ruiz J, Roache JD, Hein JM, Blount TH; STRONG STAR Consortium. Combining a stellate ganglion block with prolonged exposure therapy for posttraumatic stress disorder: A nonrandomized clinical trial. J Trauma Stress. 2022 Dec;35(6):1801-1809. doi: 10.1002/jts.22873. Epub 2022 Sep 1. PMID 36050896

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT04302181/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT04302181/ICF_001.pdf